CLINICAL TRIAL: NCT05781867
Title: Effect of Selective Manual Therapy Techniques in Chronic Obstructive Pulmonary Disease
Brief Title: Selective Manual Therapy Techniques in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira saad mohamed, M.SC physical theray, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: manual therapy in COPD
Record Dates: First submitted 2023-01-21; First posted 2023-03-23 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): 26patients will be included in this group and will receive conventional physiotherapy in form of pursed lip breathing, diaphragmatic breathing exercise and Active Range of Motion of both upper extremities
  Interventions: Other: Manual therapy and conventional physical therapy treatment
- manual therapy (Experimental): 26patients will be included in this group and will receive manual therapy (chest mobilization, diaphragmatic myofascial release, myofascial release for pectoralis minor and major, scaleni ) and conventional physiotherapy
  Interventions: Other: Manual therapy and conventional physical therapy treatment

INTERVENTIONS:
Other: Manual therapy and conventional physical therapy treatment — manual therapy (chest mobilization, diaphragmatic myofascial release, myofascial release for pectoralis minor, pectoralis major, scaleni ),pursed lip breathing, diaphragmatic breathing and active range of motion exercises of upper limbs

SUMMARY:
Our study aiming for determining the combined effect of selective manual therapy techniques in chronic obstructive pulmonary disease patients

DETAILED DESCRIPTION:
I will apply selective manual therapy techniques in form of mobilization techniques ,myofascial release techniques combined with traditional treatment to determine thier effect in chronic obstructive pulmonary disease patients

ELIGIBILITY:
Inclusion Criteria:

* All patients must diagnosed mild to moderate chronic obstructive pulmonary disease
* All patients should have foreward head and kyphosis

Exclusion Criteria:

* History of osteoporosis.
* Acute exacerbation.
* Presence of active hemoptysis
* Presence of malignant disease

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
chest expansion | pre-intervention and after 8 weeks of intervention
  caliper will be used to assess chest expansion into centimeter
(the forced vital capacity (FVC), forced expiratory volume at first second (FEV1) and FEV1/FVC will be recorded. ) | pre-intervention
  spirometry used to measure
cranio-vertebral angle and kyphotic angle in degrees | pre-intervention
  kinovea software will be used to assess in degrees
functional capacity. | pre-intervention
  Six minute walk test will be used to assess functional capacity(meter/minutes)
dyspnea score | pre-intervention
  Modified Medical Research Council dyspnea scale (mMRC dyspnea scale) will be used to assess dyspnea

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
waiting to know the results of the intervention